CLINICAL TRIAL: NCT05168605
Title: Assessing the Efficacy of Targeted Home Visits in the Management of Chronic Conditions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Nora Gimpel, Professor of Family and Community Medicine, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STU- 2019-1264
Record Dates: First submitted 2021-12-09; First posted 2021-12-23 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Hypertension; Type 2 Diabetes
MeSH Terms: conditions — Hypertension; Diabetes Mellitus, Type 2 | interventions — House Calls

STUDY DESIGN:
Intervention Model Description: This study includes prospective intervention arm and historical control arm (data will be collected via retrospective chart review).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home Visit (Experimental): Participants will receive home visit During the course of the first home visit, patients will receive routine care for diabetes and hypertension management (outcome variables are listed below) and data will be recorded in the EHR for primary outcomes. The resident physician will also assist the patient in completing enrollment in MyChart (if interested), utilizing either the resident's computer or smartphone and an internet hotspot. MyChart is a patient health platform that allows patients to contact their healthcare doctors, log health reminders, see test results, and a list of medications. The resident physician will also review a social determinants of health (SDH) screener (included in the EHR). The research faculty (licensed medical clinician) will collect blood pressure readings during this visit.
  Interventions: Other: Home visit
- Standard of care (No Intervention): Participants will receive a standard of care

INTERVENTIONS:
Other: Home visit — Patients receiving home Visits
  Arms: Home Visit

SUMMARY:
The purpose of study is to evaluate whether home visit programs are an effective method for HTN and T2DM management as compared to standard of care clinic visits.

DETAILED DESCRIPTION:
The purpose of this study is to compare the health outcomes utilizing home medical visits to manage hypertension and type 2 diabetes as compared to standard of care clinic visits.

This project has 3 overall objectives:

1. To test the efficacy of home medical visits by Family Medicine physicians specifically designed for patients with hypertension (HTN) and Type 2 Diabetes Mellitus (T2DM)
2. To compare primary outcome of the patients randomly selected for home visits to similar patients receiving usual care in the clinical setting
3. To understand the efficacy and impact of the home visit from the patient perspective

Study participant will receive usual care from a resident doctor in home. There will be (2) home visits conducted over the course of this study that will include a comprehensive assessment of hypertension, type 2 diabetes, and social factors that may be impacting their health. Study participants will also be asked to complete several questionnaires related to their knowledge of chronic diseases, personal health management, and experience of the study home visits.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ages 18-60
* Spanish or English speaking
* Diagnosis of HTN or BP >140/90 in last 3 months (based on medical record)
* Hemoglobin A1C>8 in last 6 months (based on medical record)
* Not pregnant

Exclusion Criteria:

* Current oral steroid use
* History of solid organ transplant
* Language other than English or Spanish

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-07-27 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Blood pressure | Baseline, 6 months
  Change in blood pressure will be measured at baseline, 6 months using an automated blood pressure machine. Blood pressure is measured as systolic blood pressure/diastolic blood pressure in millimeters of mercury

CONTACTS AND LOCATIONS:
Overall Officials: Nora Gimpel, M.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No